CLINICAL TRIAL: NCT05451576
Title: The Role of Sodium Selenite Supplementation in Patients With Locally Advanced Head and Neck Cancer Undergoing Concurrent Chemoradiotherapy
Brief Title: Sodium Selenite Supplementation in Patients With Head and Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, LING HANG HUONG, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 202000865A3
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Selenium; Sodium Selenite
Keywords: Sodium selenite; Selenium; chemoradiotherapy; head and neck cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium selenite (Active Comparator): 200μg/d intravenous sodium selenite was dissolved in 100 ml 0.09% NaCl run 30 minutes, will be given on day 1-5, day 8-12, day 15-19, day 22-26, day 29-33, day 36-40, day 43-47 during concurrent chemoradiotherapy.
  Interventions: Dietary Supplement: Zelnite®
- Placebo (Placebo Comparator): 100 ml intravenous 0.09% NaCl run 30 minutes, will be given on day 1-5, day 8-12, day 15-19, day 22-26, day 29-33, day 36-40, day 43-47 during concurrent chemoradiotherapy.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Zelnite® — 2pc intravenous Zelnite® will be given for 7 weeks (5 days/week).
  Arms: Sodium selenite
Dietary Supplement: Placebo — Placebo will be given for 7 weeks (5 days/week).
  Arms: Placebo

SUMMARY:
The micronutrient selenium is an essential trace element in the human body. There are more than 25 proteins in the human body contain selenium, such as glutathione peroxidase and selenoprotein, which regulate the body's antioxidant and anti-inflammatory properties. Previous literatures had shown cancer patients have lower serum selenium concentrations than normal people, and lower serum selenium levels may be associated with increased cancer mortality. More than 50% of patients with locally advanced head and neck cancer are malnourished before treatment, and these patients often have deficiency of trace elements, including selenium. In these malnourished patients, they may have to endure increased treatment toxicity and treatment interruption when receiving standard concurrent chemoradiotherapy (CCRT). Interruption of treatment may lead to reduced therapeutic efficacy and compromised survival and recurrence rate. Several small studies have investigated whether oral administration of sodium selenite in patients with head and neck cancer undergoing radiation therapy can improve side effects and affect survival rates, but the results are inconsistent. Our study will use the intravenous form of sodium selenite (Zelnite®) to investigate the effect of selenium on the treatment outcomes of locally advanced head and neck cancer patients undergoing CCRT, such as therapy-related toxicities, quality of life, changes in selenium concentration in blood, nutritional, inflammation and immune markers, and tracking long-term survival and recurrence rates.

DETAILED DESCRIPTION:
Selenium is an essential trace element for humans. It is involved in redox regulation, antioxidant functions, membrane integrity, and protection against DNA injury. In both animal models and human studies, it has been shown that selenium has cancer-protective effects and cytoprotective activities. Some mechanisms have been proposed to explain the anti-cancer effects of selenium, which include the antioxidant properties by selenoproteins, induction of conjugating enzymes that detoxify carcinogens, enhancement of the immune response, alterations in DNA methylation and blockage of the cell cycle to allow DNA repair.

There has been conflicting response regarding selenium supplementation on the reduction of toxicity, antitumor efficacy and their quality of life in patients receiving radiotherapy. In the studies by Kiremidjian-Schumacher et al. and Elango et. al, sodium selenite supplementation was shown to significantly enhance cell-mediated immune responsiveness and improve defense systems in head and neck cancer patients. Micke et al. and Zimmerman et al. demonstrated the quality of life of patients suffering from head and neck cancer with lymphedema significantly improved after selenium supplementation. In the study by Büntzel et al., selenium supplementation reduced the radiation-associated side-effects of dysphagia developments in patients with head and neck cancer patients.

However, some studies showed negative response of selenium supplementation in head and neck cancer patients. Weijl et al. showed oral selenium supplementation did not show improvement in cisplatin-induced toxicity or response rate in cancer patients. In the study by Mix et al., addition of oral selenium supplementation was well-tolerated but did not lower the incidence of severe mucositis or improve quality of life or survival outcomes in head and neck cancer patients undergoing concurrent chemoradiation (CRT). An early systematic review in Cochrane demonstrated there was still insufficient evidence to conclude efficacy of selenium in alleviating the side effects of chemotherapy or radiotherapy treatments.

The aim of this study is to investigate the effect of intravenous selenium supplementation on the treatment outcome of head and neck patients undergoing CCRT (toxicities, quality of life, overall survival, progression-free survival), selenium concentration changes during CCRT, and its correlation with nutritional, inflammation and immune markers.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven head and neck squamous cell carcinoma (oral cavity, oropharynx, hypopharynx, larynx, or metastatic cervical lymphadenopathy of unknown primary origin) who were scheduled for adjuvant or primary concurrent chemoradiotherapy (CCRT).
* American Joint Committee on Cancer 8th edition stage III, IVA, and IVB patients.
* Age 20-75 years old.
* Adequate hematopoietic or organ function (leukocyte count ≥ 3.0 x 109/L, hemoglobin ≥ 10 g/dL, platelet count ≥ 100 x109/L, serum bilirubin level ≤ 1.5 mg/dL, alanine aminotransferase (ALT) and aspartate aminotransferase levels (AST) ≤ 3 x upper limit of normal, and serum creatinine level ≤ 1.6 mg/dL or creatinine clearance ≥ 60 mL/min/1.73m2).
* ECOG performance status grade≦2.
* Subjects understand this study, agree to join this study and are able to sign the written inform consent form.

Exclusion Criteria:

* Nasopharyngeal cancer.
* History of selenium allergy or intolerance.
* Received selenium supplementation in recent 1 month.
* Uncontrolled infection - according to PI diagnosis
* Heart failure - New York Heart Association class IV
* Impaired liver function (serum total bilirubin > 2 x upper limit of normal (ULN), ALT and/or AST > 5 x ULN).
* Impaired renal function: serum creatinine > 1.5 x ULN.
* Inadequate bone marrow function (white blood cell count < 2,500 / mm3 (<2.5 x 10^9/L), platelets < 100,000 / mm3 (< 100 x 10^9/L) and hemoglobin < 10 g/dL).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Toxicities | Week 1 to Week 8
  Mucositis, pharyngitis, dermatitis, xerostomia, fatigue, infection, and cytopenia by Common Terminology Criteria for Adverse Events version 5 (CTCAE v5.0)
Pain assessment | Week 1 to Week 8
  Visual analogue scale (VAS): score ranges 0-10 (higher value indicates worse outcome)
Quality of life changes | Week 1 to Week 8
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Module (EORTC QLQ-HN43), reported in mean values (higher value indicates worse outcome)
Serum concentration changes of selenium | Week 1 to Week 8
  Serum levels of selenium during concurrent chemoradiotherapy
Changes of albumin | Week 1 to Week 12
  Serum albumin (g/dL) changes during concurrent chemoradiotherapy
Changes of transferrin | Week 1 to Week 12
  Serum transferrin (mg/dL) changes during concurrent chemoradiotherapy
Changes of total cholesterol | Week 1 to Week 12
  Total cholesterol (mg/dL) changes during concurrent chemoradiotherapy
Change of interferon-γ (IFNγ) | Week 1 to Week 8
  IFNγ (pg/mL) changes during concurrent chemoradiotherapy
Changes of tumor necrosis factor-α (TNFα) | Week 1 to Week 8
  TNFα (pg/mL) changes during concurrent chemoradiotherapy
Changes of interleukin-2 (IL-2) | Week 1 to Week 8
  IL-2 (pg/mL) changes during concurrent chemoradiotherapy
Changes of interleukin-6 (IL-6) | Week 1 to Week 8
  IL-6 (pg/mL) changes during concurrent chemoradiotherapy
Changes of granzyme B | Week 1 to Week 8
  Granzyme B (pg/mL) changes during concurrent chemoradiotherapy
Immune cells changes during concurrent chemoradiotherapy | Week 1 to Week 8
  By using Maxpar Direct Immune Profiling Assay to identify 30 subsets of immune cells

SECONDARY OUTCOMES:
Disease-free survival | 0 to 3 years
Overall survival | 0 to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hang Huong Ling, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiremidjian-Schumacher L, Roy M, Glickman R, Schneider K, Rothstein S, Cooper J, Hochster H, Kim M, Newman R. Selenium and immunocompetence in patients with head and neck cancer. Biol Trace Elem Res. 2000 Feb;73(2):97-111. doi: 10.1385/BTER:73:2:97. PMID 11049203
- [Background] Elango N, Samuel S, Chinnakkannu P. Enzymatic and non-enzymatic antioxidant status in stage (III) human oral squamous cell carcinoma and treated with radical radio therapy: influence of selenium supplementation. Clin Chim Acta. 2006 Nov;373(1-2):92-8. doi: 10.1016/j.cca.2006.05.021. Epub 2006 May 19. PMID 16831410
- [Background] Micke O, Bruns F, Mucke R, Schafer U, Glatzel M, DeVries AF, Schonekaes K, Kisters K, Buntzel J. Selenium in the treatment of radiation-associated secondary lymphedema. Int J Radiat Oncol Biol Phys. 2003 May 1;56(1):40-9. doi: 10.1016/s0360-3016(02)04390-0. PMID 12694822
- [Background] Zimmermann T, Leonhardt H, Kersting S, Albrecht S, Range U, Eckelt U. Reduction of postoperative lymphedema after oral tumor surgery with sodium selenite. Biol Trace Elem Res. 2005 Sep;106(3):193-203. doi: 10.1385/BTER:106:3:193. PMID 16141467
- [Background] Buntzel J, Riesenbeck D, Glatzel M, Berndt-Skorka R, Riedel T, Mucke R, Kisters K, Schonekaes KG, Schafer U, Bruns F, Micke O. Limited effects of selenium substitution in the prevention of radiation-associated toxicities. results of a randomized study in head and neck cancer patients. Anticancer Res. 2010 May;30(5):1829-32. PMID 20592387
- [Background] Weijl NI, Elsendoorn TJ, Lentjes EG, Hopman GD, Wipkink-Bakker A, Zwinderman AH, Cleton FJ, Osanto S. Supplementation with antioxidant micronutrients and chemotherapy-induced toxicity in cancer patients treated with cisplatin-based chemotherapy: a randomised, double-blind, placebo-controlled study. Eur J Cancer. 2004 Jul;40(11):1713-23. doi: 10.1016/j.ejca.2004.02.029. PMID 15251161
- [Background] Mix M, Singh AK, Tills M, Dibaj S, Groman A, Jaggernauth W, Rustum Y, Jameson MB. Randomized phase II trial of selenomethionine as a modulator of efficacy and toxicity of chemoradiation in squamous cell carcinoma of the head and neck. World J Clin Oncol. 2015 Oct 10;6(5):166-73. doi: 10.5306/wjco.v6.i5.166. PMID 26468453
- [Background] Dennert G, Horneber M. Selenium for alleviating the side effects of chemotherapy, radiotherapy and surgery in cancer patients. Cochrane Database Syst Rev. 2006 Jul 19;2006(3):CD005037. doi: 10.1002/14651858.CD005037.pub2. PMID 16856073